CLINICAL TRIAL: NCT04149002
Title: Improving the Clinical Encounter to Enhance Delivery of an Individualized Prematurity Prevention Plan (IP3) - The IMPaCT-IP3 Study
Brief Title: Improving the Clinical Encounter to Enhance Delivery of an Individualized Prematurity Prevention Plan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00103922
Record Dates: First submitted 2019-10-11; First posted 2019-11-04 (Actual); Results first posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Intervention Arm vs. Active Control Arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm: Weekly IP3 text messages (Other): * A narrated powerpoint presentation describing the logistical details and medical rationale for components of the IP3. Participants will view the chapters of the presentation that are relevant to their specific IP3. There are a total of 4 possible chapters (lifestyle modifications, cervix length screening/cerclage, progesterone therapy, low dose aspirin). Each chapter of the presentation is ~ 10 - 15 min in length. Each chapter also includes a 4- 5 questions pre-test and the same questions are delivered as a post-test after the presentation.
  * Print materials including a letter explaining the importance of prenatal care for preterm birth prevention to employers.
  * Text messages sent weekly to encourage the patient to continue with their IP3 and provide basic pregnancy information
  * Formal letter of encouragement from provider at 28 weeks gestation
  Interventions: Behavioral: Intervention Arm Weekly IP3 text messages
- Control Arm: General pregnancy text messages (Active Comparator): * a pre-intervention questionnaire
  * a narrated powerpoint with general information about the clinic
  * a post-presentation questionnaire
  * text messages sent approximately weekly with general pregnancy information (e.g. today your baby is about the size of an apple)
  * an exit interview
  Interventions: Other: Active Control Arm General pregnancy text messages

INTERVENTIONS:
Behavioral: Intervention Arm Weekly IP3 text messages — Subjects will be provided with a pre and post intervention survey, in addition to a narrated Powerpoint presentation focusing on the logistics of their IP3. Subjects will also receive weekly automated text messages to encourage adherence to the need for their IP3.
  Arms: Intervention Arm: Weekly IP3 text messages
Other: Active Control Arm General pregnancy text messages — Subjects will be given pre and post pre questionnaires, in addition to a narrated Powerpoint presentation about the Clinic. Subjects will also be sent weekly text messages with general pregnancy information.
  Arms: Control Arm: General pregnancy text messages

SUMMARY:
The purpose of this study is to pilot an intervention that was developed to improve uptake and adhere to an Individualized Prematurity Prevention Plan (IP3) for preterm birth prevention. Non-Hispanic Black (NHB) women are at higher risk for preterm birth compared to other racial and ethnic groups. Building on qualitative data from NHB women with input from a multidisciplinary stakeholder group, a patient-centered intervention was developed to improve uptake and adherence to an IP3 in NHB women.

DETAILED DESCRIPTION:
The study team will pilot test the intervention via a pilot randomized controlled trial. 60 pregnant NHB women will be recruited who have a history of singleton preterm birth and are currently pregnant with a singleton gestation. Consenting participants will be randomized to the intervention or an active control. The intervention includes: 1) an informational narrated powerpoint presentation that reviews the logistical details of the IP3, 2) structured encouragement via text messages and 3) employment law education sheet. The powerpoints will also be available for review on our you-tube channel for intervention patients. The active control arm includes: 1) a narrated powerpoint describing the Duke Prematurity Prevention Program and 2) text messages with general pregnancy information (i.e. it is safe to take Tylenol in pregnancy). At study intake, we will collect demographic data (age, self-described race, pregnancy history, social history, pregnancy-related anxiety scale, interpersonal processes of care and maternal social support index.

The team will collect feedback on the intervention based on an intake questionnaire and an exit interview.

Information will also be collected on adherence to the IP3 based on review of the participant's medical record. The primary aim of the study is to evaluation feasibility and acceptability. These endpoints will be measured via enrollment and participant feedback during the exit interview.

ELIGIBILITY:
Inclusion Criteria:

* self described race as Non-Hispanic Black
* history of prior singleton preterm delivery (before 37 weeks gestation)
* current singleton gestation

Exclusion Criteria:

* women with anomalous fetuses
* age below 18]
* non-English speaking

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarahn Wheeler, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Arm: Weekly IP3 Text Messages: * A narrated powerpoint presentation describing the logistical details and medical rationale for components of the IP3 (Individualized Prematurity Prevention Plan). Participants will view the chapters of the presentation that are relevant to their specific IP3. There are a total of 4 possible chapters (lifestyle modifications, cervix length screening/cerclage, progesterone therapy, low dose aspirin). Each chapter of the presentation is ~ 10 - 15 min in length. Each chapter also includes a 4- 5 questions pre-test and the same questions are delivered as a post-test after the presentation.
  * Print materials including a letter explaining the importance of prenatal care for preterm birth prevention to employers.
  * Text messages sent weekly to encourage the patient to continue with their IP3 and provide basic pregnancy information
  * Formal letter of encouragement from provider at 28 weeks gestation
  Intervention Arm Weekly IP3 text messages: Subjects will be provided with a pre and post intervention survey, in addition to a narrated Powerpoint presentation focusing on the logistics of their IP3. Subjects will also receive weekly automated text messages to encourage adherence to the need for their IP3.
- Control Arm: General Pregnancy Text Messages: * a pre-intervention questionnaire
  * a narrated powerpoint with general information about the clinic
  * a post-presentation questionnaire
  * text messages sent approximately weekly with general pregnancy information (e.g. today your baby is about the size of an apple)
  * an exit interview
  Active Control Arm General pregnancy text messages: Subjects will be given pre and post pre questionnaires, in addition to a narrated Powerpoint presentation about the Clinic. Subjects will also be sent weekly text messages with general pregnancy information.
Period: Overall Study
Arm/Group | Intervention Arm: Weekly IP3 Text Messages | Control Arm: General Pregnancy Text Messages
Started | 14 | 16
Completed | 12 | 16
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention Arm: Weekly IP3 Text Messages: * A narrated powerpoint presentation describing the logistical details and medical rationale for components of the IP3. Participants will view the chapters of the presentation that are relevant to their specific IP3. There are a total of 4 possible chapters (lifestyle modifications, cervix length screening/cerclage, progesterone therapy, low dose aspirin). Each chapter of the presentation is ~ 10 - 15 min in length. Each chapter also includes a 4- 5 questions pre-test and the same questions are delivered as a post-test after the presentation.
  * Print materials including a letter explaining the importance of prenatal care for preterm birth prevention to employers.
  * Text messages sent weekly to encourage the patient to continue with their IP3 and provide basic pregnancy information
  * Formal letter of encouragement from provider at 28 weeks gestation
  Intervention Arm Weekly IP3 text messages: Subjects will be provided with a pre and post intervention survey, in addition to a narrated Powerpoint presentation focusing on the logistics of their IP3. Subjects will also receive weekly automated text messages to encourage adherence to the need for their IP3.
- Total: Total of all reporting groups
Arm/Group | Intervention Arm: Weekly IP3 Text Messages | Control Arm: General Pregnancy Text Messages | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.9 (5.3) | 32.1 (7.0) | 31.5 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 16 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 16 | 30
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Measured by Number of Recruited Eligible Patients Enrolled
Description: Enrollment target of 30% of eligible patients recruited.
Time Frame: study duration (approximately 14 months)
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Patients Recruited: Patients who met all study inclusion criteria.
Arm/Group | Eligible Patients Recruited
Number analyzed (Participants) | 54
Participants | 30

2. Primary Outcome: Acceptability as Measured by Number of Participants Who Completed the Study
Description: Completion target of 80% participants retained in study protocol.
Time Frame: study duration (approximately 14 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm: Weekly IP3 Text Messages | Control Arm: General Pregnancy Text Messages
Number analyzed (Participants) | 14 | 16
Participants | 12 | 16

3. Secondary Outcome: IP3 Adherence as Measured by Number of Participants With Patient and EMR (Electronic Medical Record) Report of Medication Compliance
Time Frame: approximately 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm: Weekly IP3 Text Messages | Control Arm: General Pregnancy Text Messages
Number analyzed (Participants) | 14 | 16
Participants | 1 | 3

4. Secondary Outcome: Pregnancy Specific Anxiety (PSA)
Description: Pregnancy specific anxiety is a 4-question scale. Each question can be answered on a range of 1 to 5. Scores were averaged to produce one mean PSA score ranging from 1-5. Higher scores are negative and denote increased anxiety.
Time Frame: baseline, 28 weeks
Population: Participants who completed the PSA questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm: Weekly IP3 Text Messages | Control Arm: General Pregnancy Text Messages
Number analyzed (Participants) | 11 | 15
score on a scale
  Baseline | 2.6 (1.0) | 2.4 (0.9)
  28 Weeks | 2.3 (0.9) | 2.3 (0.6)

5. Secondary Outcome: Interpersonal Process of Care (IPC-18) at Protocol Completion - Communication Domain
Description: The IPC is an 18-question questionnaire that asks participants about their experience with receiving care within a specific clinic (in this case the Duke Perinatal Durham Clinic). All IPC items use an identical set of response options: 1='never'; 2='rarely'; 3='sometimes'; 4='usually'; 5='always.' Item responses are averaged, not summed; thus, scores have a possible range of 1-5. All scales are scored so that higher scores indicate higher frequency of the labeled interpersonal process: Lack of clarity (higher scores are negative), Elicits concern (higher scores are positive), and Explain results (higher scores are positive).
Time Frame: protocol completion (approximately 1 year)
Population: Participants who completed the IPC-18 questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm: Weekly IP3 Text Messages | Control Arm: General Pregnancy Text Messages
Number analyzed (Participants) | 11 | 15
score on a scale
  Lack of clarity | 1.6 (0.6) | 1.6 (1.1)
  Elicits concern | 4.6 (0.6) | 4.7 (0.6)
  Explain results | 4.5 (0.6) | 4.6 (0.7)

6. Secondary Outcome: Interpersonal Process of Care (IPC-18) at Protocol Completion - Decision Making Domain
Description: The IPC is an 18-question questionnaire that asks participants about their experience with receiving care within a specific clinic (in this case the Duke Perinatal Durham Clinic). All IPC items use an identical set of response options: 1='never'; 2='rarely'; 3='sometimes'; 4='usually'; 5='always.' Item responses are averaged, not summed; thus, scores have a possible range of 1-5. All scales are scored so that higher scores indicate higher frequency of the labeled interpersonal process: Decision Making (higher scores are positive, denoting more collaborative decision making between the clinician and patient).
Time Frame: protocol completion (approximately 1 year)
Population: Participants who completed the IPC-18 questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm: Weekly IP3 Text Messages | Control Arm: General Pregnancy Text Messages
Number analyzed (Participants) | 11 | 15
score on a scale | 4.4 (1.1) | 4.8 (0.4)

7. Secondary Outcome: Interpersonal Process of Care (IPC-18) at Protocol Completion - Interpersonal Style Domain
Description: The IPC is an 18-question questionnaire that asks participants about their experience with receiving care within a specific clinic (in this case the Duke Perinatal Durham Clinic). All IPC items use an identical set of response options: 1='never'; 2='rarely'; 3='sometimes'; 4='usually'; 5='always.' Item responses are averaged, not summed; thus, scores have a possible range of 1-5. All scales are scored so that higher scores indicate higher frequency of the labeled interpersonal process: Emotional support (higher scores are positive), Discrimination due to race/ethnicity (higher scores are negative), Disrespectful to office staff (higher scores are negative).
Time Frame: protocol completion (approximately 1 year)
Population: Participants who completed the IPC-18 questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm: Weekly IP3 Text Messages | Control Arm: General Pregnancy Text Messages
Number analyzed (Participants) | 11 | 15
score on a scale
  Emotional support | 4.7 (0.5) | 4.8 (0.4)
  Discrimination due to race/ethnicity | 1.5 (0.7) | 1.3 (0.8)
  Disrespectful to office staff | 1.2 (0.3) | 1.1 (0.5)

8. Secondary Outcome: Change in Maternal Social Support Scale (MSSS)
Description: The MSSS is a six-question scale that quantifies a pregnant woman's social support. Social factors (lack of family support, low friendship network, lack of help from spouse/partner, conflict with spouse/partner, feeling controlled by spouse/partner, and feeling unloved by spouse/partner) are combined in a 6-item self-report 5-point Likert scale. The total possible score for the scale is between 6 and 30, with higher scores indicating increased support.
Time Frame: baseline to protocol completion (approximately 1 year)
Population: Participants who completed the MSSS questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm: Weekly IP3 Text Messages | Control Arm: General Pregnancy Text Messages
Number analyzed (Participants) | 11 | 15
score on a scale | 0.1 (1.5) | -1.4 (2.4)

9. Secondary Outcome: Gestational Age at Delivery in Weeks
Time Frame: approximately 40 weeks
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Intervention Arm: Weekly IP3 Text Messages | Control Arm: General Pregnancy Text Messages
Number analyzed (Participants) | 14 | 16
weeks | 34.0 (6.1) | 35.7 (3.5)

10. Secondary Outcome: Birth Weight in Grams
Time Frame: approximately 40 weeks
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Intervention Arm: Weekly IP3 Text Messages | Control Arm: General Pregnancy Text Messages
Number analyzed (Participants) | 14 | 16
grams | 2442.5 (1255.9) | 2607.9 (750.6)

11. Secondary Outcome: Number of Neonates Admitted to the Newborn Intensive Care Unit (NICU)
Time Frame: approximately 40 weeks
Measure: Count of Units; unit: Neonates
Units Other Than Participants: Neonates
Arm/Group | Intervention Arm: Weekly IP3 Text Messages | Control Arm: General Pregnancy Text Messages
Number analyzed (Participants) | 14 | 16
Number analyzed (Neonates) | 14 | 16
Neonates | 5 | 4

12. Secondary Outcome: Length of Delivery Hospital Admission in Days
Time Frame: approximately 40 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Intervention Arm: Weekly IP3 Text Messages | Control Arm: General Pregnancy Text Messages
Number analyzed (Participants) | 14 | 16
days | 2 [2 to 3] | 3 [2 to 3]

ADVERSE EVENTS:
Time Frame: Approximately 1 year
Description: Adverse Events are for Mothers only.
Arm/Group | Intervention Arm: Weekly IP3 Text Messages | Control Arm: General Pregnancy Text Messages
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 0/14 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT04149002/Prot_SAP_001.pdf
  • Informed Consent Form (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/02/NCT04149002/ICF_000.pdf